CLINICAL TRIAL: NCT03079453
Title: An Approach to Reduce Uvula Edema After Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Nazan Degirmenci, MD, Bezmialem Vakif University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 11/18-03.06.2015
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Edema
Keywords: Dexamethasone; Tonsillectomy; Uvula; Edema; Uvula edema; Post-tonsillectomy
MeSH Terms: conditions — Edema | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Thirty patients ages 18 to 48 years who underwent tonsillectomy included in this prospective randomized clinical trial. The patients in Group 1 (n:15) were injected with dexamethasone (1 ml, 8 mg) through the uvula and soft palate tissue directly at three points (three points on the connection of the uvula, and palatum molle) before tonsillectomy. Group 2 (n:15) patients had tonsillectomy without dexamethasone injection.Blinded observers made examinations of the groups postoperative on the first and fifth days and evaluated the uvula edema by using the uvula edema scale that the investigators developed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): The patients in Group 1 (n:15) were injected with dexamethasone (1 ml, 8 mg) through the uvula and soft palate tissue directly at three points (three points on the connection of the uvula, and palatum molle) before tonsillectomy .
  Interventions: Drug: Dexamethasone
- Group 2 (No Intervention): Group 2 (n:15) patients had tonsillectomy without dexamethasone injection.

INTERVENTIONS:
Drug: Dexamethasone — The patients in Group 1 were injected with dexamethasone (1 ml, 8 mg) through the uvula and soft palate tissue directly before tonsillectomy
  Other Names: Dexasone
  Arms: Group 1

SUMMARY:
A prospective randomized clinical trial that included thirty subjects who underwent tonsillectomy. The patients in Group 1 (n:15) were injected with dexamethasone (1 ml, 8 mg) through the uvula and soft palate tissue directly before tonsillectomy. Group 2 (n:15) patients had tonsillectomy without dexamethasone injection. Patients were examined preoperatively and postoperative on the first and fifth days. In this study investigators tried an approach of dexamethasone application to reduce uvula edema after tonsillectomy.

DETAILED DESCRIPTION:
Thirty patients between the ages of 18 and 48 years were enrolled in this prospective randomized clinical trial from July 2015 to July 2016. The study was carried out in a tertiary referral center in Istanbul, Turkey. Permission for the study was obtained from Bezmialem Vakif University Clinical Research Ethics Committee, on 03 June 2015, number11/18.

The patients in Group 1 (n:15) were injected with dexamethasone (1 ml, 8 mg) through the uvula and soft palate tissue directly at three points (three points on the connection of the uvula, and palatum molle) before tonsillectomy. Group 2 (n:15) patients had tonsillectomy without dexamethasone injection. All patients had the operation under general anesthesia by utilizing the same protocol. Both of the groups were not given iv/im dexamethasone perioperatively. The surgical technique for tonsillectomy was bipolar cautery dissection performed by the same surgeon. The oropharyngeal area was examined and photographed endoscopically preoperatively and postoperative on the first and fifth days. All of the participants were examined with an 8mm diameter 70º endoscope. The photographs of the oropharynx (anterior plicas, tonsils, uvula, posterior oropharynx) were taken by holding the endoscope positioned vertically to the mouth. Blinded observers made examinations of the groups at the postoperative first and fifth days and evaluated the uvula edema by using the uvula edema scale that the investigators developed.

The investigators used a scale for grading uvula edema. There is no such scale in the English literature so the investigators developed a scale for grading uvula edema. The investigators grade edema from 1 to 5 as an increase of the edema area. It is called Grade 1 if there was elongation only at the tip of the uvula. If there was edema in the body and base of the uvula, it is called Grade 2. If the uvula edema was spread over a larger area than Grade 2, and if there was involvement in the unilateral plica, it is called Grade 3. If it was spread to both pharyngeal plicas, it is called grade 4. If the uvula edema caused the complete blockage of the posterior pharyngeal tract, it is called Grade 5.

The statistical tests were conducted using the Statistical Package for the Social Sciences version 24.0 for Windows (SPSS Inc., Chicago, Illinois, USA). All quantitative variables were estimated using measures of central location (i.e., mean and median) and measures of dispersion (i.e., standard deviation [SD]). Data normality was tested using the Shapiro-Wilk tests of normality. Descriptive statistical analysis were made. Paired t test was used for comparison of intra-group quantitative data. Independent t test was used to compare groups of quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with recurrent tonsillitis but no sleep apnea
* Subjects older than eighteen years old
* Subjects were planned to have only tonsillectomy procedure

Exclusion Criteria:

* Subjects who must have additional procedures other than tonsillectomy
* Subjects younger than eighteen years old
* Subjects that had intravenous dexamethasone administration perioperatively

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of local dexamethasone administration to reduce uvula edema after tonsillectomy evaluated by using the uvula edema scale | Postoperative first and fifth days
  Uvula edema wase evaluated at the postoperative first and fifth days by using the uvula edema scale that the investigators developed.

CONTACTS AND LOCATIONS:
Overall Officials: Selahattin Tugrul, Assoc. Prof., Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No